CLINICAL TRIAL: NCT02290743
Title: The Effect of One Application of Kinesio Tape on Muscle Strength in Quadriceps Femoris on Patients With Knee Problems or Pain and Weak Quadriceps Femoris - a Randomized Controlled Trial
Brief Title: Effect of Kinesio Taping on Muscle Strength in Quadriceps Femoris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Nina Paulsen, Physiotherapist and masterstudent in Sports Physiotherapy, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KT-QF
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Anterior Knee Pain; Muscle Weakness; Knee Symptoms
MeSH Terms: conditions — Muscle Weakness | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinesio tape (Experimental): Kinesio tape on quadriceps femoris
  Interventions: Other: Kinesio tape
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Kinesio tape — Application of one Kinesio tape with 0-30 % tension over the muscle fibers of the quadriceps femoris in a stretched position. The tape can be divided into several tails to cover the whole muscle from origin to insertion.
  Other Names: Kinesio taping; Kinesio tex taping
  Arms: Kinesio tape

SUMMARY:
The purpose of this project is to investigate the effect of Kinesio tape on muscle strength of the quadriceps femoris in people with knee pain or symptoms and decreased muscle strength in the quadriceps femoris - a randomized controlled trial.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of recoil tape with 0-30% tension, by using one application of Kinesio tape over the muscle fibers of the quadriceps femoris from its origin to its insertion. The participants will be divided into intervention group (taping) and control group (no intervention). Muscle strength test will be performed before and immediately after taping (20-30 minutes) for both groups using hand-held dynamometer measurements (MicroFET 3).

Work is based on the following hypothesis: "Kinesio taping using recoil taping provides increased isometric muscle strength in quadriceps femoris immediately after application".

ELIGIBILITY:
Inclusion Criteria:

* Shoulder problems
* Low muscle strength in quadriceps femoris
* Positive manual recoil-test for the quadriceps femoris

Exclusion Criteria:

* Knee surgery <3 month
* Pathology in the knee related to tumors, fractures, neurology, rupture of tendons

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 30 minutes
  Maximal isometric muscle strength monitored by a hand-held dynamometer (microFET 3)

SECONDARY OUTCOMES:
Time of break force | 30 minutes
  How long the patient can hold against the pressure from the investigator until the force breaks
Self-reported strength - effort scale | 30 minutes
  Self-reported muscle strength from 0-10 (0 is nothing, 1 is extremely weak and 10 is extremely strong)

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Myklebust, Phd, PT, Study Director — Department of Sports Medicine
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Oslo County, Norway